CLINICAL TRIAL: NCT02529969
Title: Curcumin Supplementation and Type 2 Diabetes
Brief Title: Effects of Curcumin Supplementation on Lipid Profile and Inflammatory Markers of Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 615
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Non Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- intervention (Active Comparator): 500 mg curcumin capsule
  Interventions: Dietary Supplement: curcumin
- placebo (Placebo Comparator): 500 mg placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: curcumin
  Arms: intervention
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
Diabetes mellitus is the most common endocrine disorder, causes many complications such as micro- and macro-vascular diseases. Various kinds of antidiabetic drugs have been developed, but most of them have side effects. Recently, the use of natural plant products has gained more attention among scientists in order to prevent diabetic vascular complications. Curcumin is a natural yellow product derived from the turmeric rhizome which has shown to be non-toxic and exhibits various bio¬logical activities such as anti-oxidant, anti-inflammatory, anti-carcinogenic, and anti-diabetic effects. Curcumin is effective in reducing glycemic index and hyperlipidemia in rodent models and is relatively inexpensive and safe. Most of the studies conducted on animal model, and just a few of them are on human model. The present study was planned to evaluate the effects of curcumin supplementation on serum levels of lipid profile and inflammatory markers in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. Tendency to participate
2. Age range of 40-65
3. Suffering from diabetes type 2 ( between 1 to 10 yeares)
4. BMI 18/5-30
5. Patients with diabetes who administer oral hypoglycemic agents and do not use

Exclusion Criteria:

1. patients with liver diseases
2. patients with kidney diseases
3. patients with inflammatory diseases
4. patients with liver diseases
5. Administering herbal agents
6. Administering multivitamins and minerals in past 3 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Triglyceride | 12 weeks

SECONDARY OUTCOMES:
C-Reactive Protein | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran